CLINICAL TRIAL: NCT04965909
Title: Online Pain Neuroscience Education and Graded Exposure to Movement in Breast Cancer Survivors: Protocol of a Randomised Controlled Trial.
Brief Title: Pain Neuroscience Education and Graded Exposure to Movement in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Patricia Martínez Miranda, Doctoranda Programa del Doctorado Interuniversitario en CCSS, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0379520202023
Record Dates: First submitted 2021-06-26; First posted 2021-07-16 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Breast Neoplasms; Pain, Chronic; Quality of Life
Keywords: breast cancer; pain; quality of life; pain neuroscience education; graded exposure to movement; therapeutic exercise
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Clinical Trial of two groups (experimental and control) will be carried out.
Who Masked: Investigator, Outcomes Assessor
Masking Description: double-blind (researcher and statistician)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational and therapeutic exercise program (Experimental): Participants will receive a 3-month online physiotherapy program comprised of 'pain neuroscience education' (month 1) and 'gradual exposure to movement' (month 2 and 3). They will receive an informative booklet online.
  Interventions: Other: Online physiotherapy protocol based on pain neuroscience education and gradual exposure to movement.
- Passive control group (usual care) (No Intervention): Participants will receive the 'usual care'. They will receive an informative booklet online and the possibility of receiving the therapeutic program, once the study is completed.

INTERVENTIONS:
Other: Online physiotherapy protocol based on pain neuroscience education and gradual exposure to movement. — Online group therapeutic program (small groups), applied for 3 months.
  Arms: Educational and therapeutic exercise program

SUMMARY:
Introduction: Pain stands out among the sequelae that affect the quality of life of breast cancer survivors. Pain neuroscience education and graded exposure to movement are therapeutic approaches that have been shown to be effective in the management of chronic pain in other populations. However, there are no previous studies that combine them in this population. Objective: To evaluate the effectiveness of an online physiotherapy focused-person program which combines pain neuroscience education and graded exposure to movement, to improve the quality of life of breast cancer survivors. Methodology: The design of the study is a randomised controlled clinical trial and the sample will be 40 breast cancer survivors with pain in the last 6 months. A random method will be used to assign participants into two groups (experimental and control). The evaluator and statistician will be blinded to participant allocation while the experimental group will receive the therapeutic program which combines pain neuroscience education and graded exposure to movement-based intervention throughout therapeutic yoga; the control will be a passive group. There will be four points of assessment: the main outcome assessed will be quality of life measured by the Functional Assessment of Cancer Therapy - Breast (FACT-B+4) and the secondary outcomes are variables related to pain experience (catastrophising, self-efficacy, kinesiophobia and fear-avoidance behaviours). All will be assessed using validated methods. SPSS program will be used for the data analysis. A mixed-model analyses of variance ANOVA (2x4) will be used to study the effects of the treatment on the dependent variables. An intention-to-treat analysis will be performed. All statistical tests will be performed considering a confidence interval of 95%. Trial record: NCT04965909.

DETAILED DESCRIPTION:
Study Design A randomised controlled clinical trial will be carried out according to the Consolidated Standards of Reporting Trials (CONSORT) Statement for its development. In addition, the Template for Intervention, Description and Replication Checklist (TIDieR) will be used as a guide to provide transparency and make the intervention replicable. Also, the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) was followed to develop this protocol. The protocol of this study has been registered on clinicaltrials.org with the registry number: NCT04965909.

Sampling method and sample's size calculation For sampling, non-probabilistic convenience and snowball methods will be used. Sample size was calculated using the G*Power software, version 3.1.9.7 (Heinrich-Heine University, Düsseldorf, Germany), and considering the previous data reported by Park et al., (2012) for the variable global Quality of life (Functional Assessment of Cancer Therapy - Breast, FACT-B). We considered 2 groups and 4 measurements, a type I risk or α 0.05, type II risk or β 0.20 (study power of 80%), and a partial Eta2 effect size of 0.049. This generated a sample of 40 individuals, including an estimated 15% dropout rate. Figure 1 shows the study flow diagram.

Subjects' recruitment The sample for this study will be recruited through the dissemination of the project using social networks and with the collaboration of three Spanish breast carcer survivor support associations (Amama Sevilla, AGAMAMA and ASAMMA). Participation in the study will be voluntary. All participants will be facilitated by written informed consent that must be signed to be part of the clinical trial.

Group assignment and masking This study will have two groups (experimental and control). For assignment, a random method will be carried out using an online tool called 'random allocation software'. A stratified allocation was applied according to the women's age (≤45 years old or >45 years old). On each of the strata, a randomisation will be carried out by blocks of constant size. The assignment sequence will be hidden from the evaluator and the study subjects through an automated assignment system. The preparation of the sequence, the inclusion of the individuals in each group and the assignment of the treatments will be carried out by different members of the research team. On the other hand, the evaluator and statistician will be blinded. Nonetheless, the therapist and subject will not be able to be blinded because of the type of intervention.

Assessment points, method of data collection and outcomes The outcomes will be assessed at four points during the entire study period: before the intervention (T0), after the experimental group completes the first part of the intervention based on PNE (T1), after complete intervention (T2) and at the 3-month follow-up (T3) (Figure 2).

All data will be collected in a format model. All data were encrypted and only members of the research team will have access to the data of the participants. The outcomes will be assessed using validated scales or questionnaires that women will complete by themselves. In addition, extra information related to their pain context will be collected by two evaluators in an online meeting. The evaluators will have previous experience in the issue and will be trained before the interviews.

The main outcome of this trial is quality of life measured by The Functional Assessment of Cancer Therapy - Breast (FACT-B+4). In addition, five secondary outcomes related to health will be measured: intensity of pain using the Brief Pain Inventory - Short Form (BPI-SF), catastrophising level using the Pain Catastrophising Scale, self-efficacy level using the Pain Self-efficacy questionnaire (PSEQ), Kinesiophobia using the Tampa Scale for Kinesiophobia (TSK-11) and fear-avoidance behaviours using the Fear Avoidance Components Scale Questionnaire - Spanish Version (FACS-SP).

Method for results and data analysis For the data analysis, a data matrix will be prepared according to the coding methods that have been described in the outcomes section. A descriptive and inferential statistical analysis will be carried out, assuming that the groups are independent. The SPSS program, version 26.0 for Windows will be used for data analysis.

First, the Shapiro-Wilk test will be used to determine whether there is a normal distribution. Then, a descriptive analysis of the data will be conducted. The absolute count and percentages of each category will be calculated in the nominal qualitative variables. For the quantitative variables adjusted to the normality, the mean and standard deviation will be provided, while the median and the first and third quartiles will be provided in those that are not adjusted to normality. Next, the homogeneity in the baseline between the experimental and control groups will be studied with respect to the sociodemographic and clinical variables and pre-test of all dependent variables. In the dichotomous nominal qualitative variables, Pearson's bilateral asymptotic Chi2 test will be used, or, failing that, Fisher's exact test. In the polytomous nominal qualitative variables, Pearson's bilateral asymptotic Chi2 test or Pearson's exact test will be used. On the other hand, in the quantitative variables adjusted to normality that are homoscedastic, we will use the student's t test for independent samples and the Welch t test in those that are heteroscedastic. In quantitative variables that do not adjust to normality, the Mann-Whitney U test will be used. On the other hand, in those variables in which the 4 measurements are adjusted to normality in both intervention groups, a mixed-model analyses of variance factorial ANOVA (2x4) will be used to study the effects of the treatment on the dependent variables evaluated in the present investigation, considering the group as a between-subject factor and time (the different measurements performed) as a within-subject factor. The hypothesis of interest will be the interaction group by time with an a priori alpha level of 0.05. In addition, the effect size of the observed differences will be estimated by calculating the partial Eta squared coefficient. In those variables in which none of the measurements in either of the two intervention groups adjust to normality, the following analyses will be implemented: the measurements made of the intragroup dependent variables will be compared (considering each of the intervention groups in isolation). In those variables in which all of the measurements are normal in one of the two intervention groups, we will use the ANOVA test of repeated measures. If any of the measurements do not adjust to normality, we will use the Friedman ANOVA test. Next, to compare the inter-group dependent variables, the difference between the value of each pair of measurements will be calculated for each dependent variable, calling such values "differences". In addition, the percentages of change in the scores between each pair of measurements were established. Finally, the values obtained in the "differences in scores" and in the "percentage changes in scores" in the two groups will be compared. For this we use Student's t test for independent samples, in the differences and percentages of change that are normal and homoscedastic, while in the normal and heteroscedastic we will use the Welch t test. The effect size was estimated by calculating Cohen's d coefficient. In the event that such differences are not normal, we will used the Mann-Whitney U test and the effect size will be found by calculating Rosenthal's r with the formula: r=Z/√N. An "intention to treat" analysis will be performed in the study of the effects of the applied intervention. All statistical tests will be performed considering a confidence interval (hereinafter CI) of 95% (p-value <0.05).

Planned timing The project would be carried out from 2020 to 2024.

Ethical considerations For the preparation of this study, all relevant ethical considerations have been made. In addition, this program has the approval of the Research Ethics Committee (CEI) of the Virgen Macarena - Virgen del Rocío University Hospitals.

In accordance with Organic Law 3/2018, of December 5, on the Protection of Personal Data and guarantee of digital rights and prior verbal and written information, this study will have the express written consent of each participant. This will be delivered together with the informed consent revocation sheet. All personal data will be treated properly, not being disclosed under any circumstances and not being misused.

ELIGIBILITY:
Inclusion criteria:

* Woman aged between 18 - 65 years.
* Diagnosis of stage 0 - III breast cancer.
* Primary treatment (surgery, radiotherapy and chemotherapy) completed at least 3 months ago may still be receiving hormonal therapy.
* Pain related to primary treatment in the last 6 months.
* Access to Internet and an electronic device that allows the use of the applications used in this study and skills for their use or assistance from a close person who has them.
* Ability to communicate fluently verbally and in writing in the language of the research team (Spanish).
* Approval of participation in the study by the coordinator of the health team that assisted her during the course of cancer and its treatment.

Exclusion criteria:

* Another previous type of cancer or breast cancer recurrence in a period of less than 1 year.
* Medical diagnosis of a neurological, autoimmune or cardiovascular disease.
* Some type of pathology that is associated with a contraindication to physical exercise.
* Diagnosis of serious psychiatric or neurologic disorders that do not allow the participant to follow orders.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from quality of life | Four evaluations will be made, before the intervention (T0, at the baseline), at the end of the application of PNE module (T1, 1 month), at the end of the GEM intervention (T2, 3 month) and at 3 months of follow-up (T3).
  Quality of life measured by the Functional Assessment of Cancer Therapy - Breast (FACT-B+4). The FACT-B+4 is a 41-item instrument designed to measure six domains of QOL in breast cancer patients: Physical, social, emotional and functional well-being, and breast-cancer (BCS) and lymphedema (ARM) subscales. The score obtained ranges from 0-148 points. The ARM subscale was not included in the total score. A higher score translates into a better quality of life.

SECONDARY OUTCOMES:
Change from pain intensity | Four evaluations will be made, before the intervention (T0, at the baseline), at the end of the application of PNE module (T1, 1 month), at the end of the GEM intervention (T2, 3 month) and at 3 months of follow-up (T3).
  Pain intensity measured by the Brief Pain Inventory - Short Form (BPI - SF). The PBI -SF is a 9-item instrument designed to measure pain intensity and pain interference with the diary daily activities. The questionnaire has two subareas, one related to pain intensity, whose score ranges from 0-50, with a higher score being an indication of greater intensity; and another related to the interference of pain in activities of daily living, whose score ranges from 0-70, with a higher score being indicative of a greater impact on daily life.
Change from catastrophism level | Four evaluations will be made, before the intervention (T0, at the baseline), at the end of the application of PNE module (T1, 1 month), at the end of the GEM intervention (T2, 3 month) and at 3 months of follow-up (T3).
  Catastrophim level measured by the Pain Catastrophizing Scale. This scale allows us to assess the degree of catastrophizing of pain in adolescents and adults who face this condition as a result of various pathologies or diseases. The scale consists of 3 subscales (rumination, magnification and helplessness), whose items will be valued from 0 (nothing) to 4 (all the time) to obtain a total score that ranges between 0-52. A higher score translates into a higher level of catastrophizing.
Change from self-efficacy level | Four evaluations will be made, before the intervention (T0, at the baseline), at the end of the application of PNE module (T1, 1 month), at the end of the GEM intervention (T2, 3 month) and at 3 months of follow-up (T3).
  Self-efficacy level measured by the pain self-efficacy questionnaire (PSEQ). The PSEQ is a 22-item instrument designed to measure self-efficacy level. Each item is scored from 0 - 10. 0 is equal to 'I think I am totally incapable' and 10 is equal to 'I think I am totally capable'. The total score ranges from 0-220. A higher score on the questionnaire corresponds to a higher level of self-efficacy.
Change from Kinesiophobia | Four evaluations will be made, before the intervention (T0, at the baseline), at the end of the application of PNE module (T1, 1 month), at the end of the GEM intervention (T2, 3 month) and at 3 months of follow-up (T3).
  Kinesiophobia measured by the Tampa Scale for Kinesiophobia (TSK-11). This scale is one of the most used to evaluate kinesiophobia in patients with pain. It is composed of two factors (avoidance of activity and harm) with a total of 11 items that are valued from 1 (totally disagree) to 4 (totally agree). The total score obtained ranges from 11 - 44. More punctuation shows higher kinesiophobia level.
Change from Fear Avoidance Beliefs | Four evaluations will be made, before the intervention (T0, at the baseline), at the end of the application of PNE module (T1, 1 month), at the end of the GEM intervention (T2, 3 month) and at 3 months of follow-up (T3).
  Fear avoidance beliefs measured by the Fear Avoidance Components Scale Questionnaire - Spanish Version (FACS - SP) . The FACS- SP is a questionnaire that allows us to evaluate patient's fear of pain and consequent avoidance of physical activity due to fear. The questionnaire consists of 20 items in which a patient rates his agreement with each statement on a 6-point Likert scale. Where 0 = completely disagree, 6 = completely agree. There is a maximum score of 100. A higher score indicates more strongly held fear-avoidance beliefs. Five severity levels are available for clinical interpretation: subclinical (0-20), mild (21-40), moderate (41-60), severe (61-80), and extreme (81-100).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Sevilla, departamento de Fisioterapia, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
The personal data of the participants will be treated in accordance with the Organic Law 3/2018, of December 5, on the Protection of Personal Data and guarantee of digital rights

REFERENCES:
- [Background] Watson JA, Ryan CG, Cooper L, Ellington D, Whittle R, Lavender M, Dixon J, Atkinson G, Cooper K, Martin DJ. Pain Neuroscience Education for Adults With Chronic Musculoskeletal Pain: A Mixed-Methods Systematic Review and Meta-Analysis. J Pain. 2019 Oct;20(10):1140.e1-1140.e22. doi: 10.1016/j.jpain.2019.02.011. Epub 2019 Mar 1. PMID 30831273
- [Background] De Groef A, Penen F, Dams L, Van der Gucht E, Nijs J, Meeus M. Best-Evidence Rehabilitation for Chronic Pain Part 2: Pain during and after Cancer Treatment. J Clin Med. 2019 Jul 5;8(7):979. doi: 10.3390/jcm8070979. PMID 31284377
- [Background] Cramer H, Lauche R, Klose P, Lange S, Langhorst J, Dobos GJ. Yoga for improving health-related quality of life, mental health and cancer-related symptoms in women diagnosed with breast cancer. Cochrane Database Syst Rev. 2017 Jan 3;1(1):CD010802. doi: 10.1002/14651858.CD010802.pub2. PMID 28045199
- [Background] Gatchel RJ, Peng YB, Peters ML, Fuchs PN, Turk DC. The biopsychosocial approach to chronic pain: scientific advances and future directions. Psychol Bull. 2007 Jul;133(4):581-624. doi: 10.1037/0033-2909.133.4.581. PMID 17592957
- [Derived] Martinez-Miranda P, Jimenez-Rejano JJ, Munoz-Fernandez MJ, Garcia-Munoz C, Casuso-Holgado MJ. Effectiveness of an interactive online group intervention based on pain neuroscience education and graded exposure to movement in breast cancer survivors with chronic pain: a randomised controlled trial. Support Care Cancer. 2024 Oct 7;32(10):705. doi: 10.1007/s00520-024-08887-4. PMID 39373766
- [Derived] Martinez-Miranda P, Casuso-Holgado MJ, Garcia-Munoz C, Munoz-Fernandez MJ, Jimenez-Rejano JJ. Online pain neuroscience education and graded exposure to movement in breast cancer survivors: protocol of a randomized controlled trial. Front Med (Lausanne). 2024 Feb 28;11:1355964. doi: 10.3389/fmed.2024.1355964. eCollection 2024. PMID 38482528